CLINICAL TRIAL: NCT05746988
Title: Carrageenan for the Prevention of Oral HPV Infection: a Feasibility, Randomized Clinical Trial
Brief Title: Carrageenan for the Prevention of Oral HPV Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dr. Belinda Nicolau, Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A03-M01-22A
Record Dates: First submitted 2023-01-17; First posted 2023-02-28 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Human Papilloma Virus
Keywords: Oral HPV infection; Mouthwash; Carrageenan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carrageenan-based Mouthwash (Experimental): Mouthwash with Carrageenan as an active ingredient
  Interventions: Other: Mouthwash gargling
- Placebo Mouthwash (Placebo Comparator): Mouthwash without Carrageenan but similar in colour, taste, and "mouthfeel" to the experimental mouthwash
  Interventions: Other: Mouthwash gargling

INTERVENTIONS:
Other: Mouthwash gargling — 15 - 20 ml of mouthwash to be gargled vigorously for 30 to 60 seconds daily (morning and night) as an adjunct to regular toothbrushing, and before and/or immediately after sexual activities.

SUMMARY:
This is a placebo-controlled, triple-blind randomized clinical trial (RCT) designed to evaluate the feasibility of conducting a larger multicentric RCT investigating the effect of a Carrageenan mouthwash on oral HPV infection. Eligible participants will complete a single in-person visit at baseline, filling out a questionnaire on their electronic device and giving an oral rinse sample for HPV testing. They will receive an adequate supply of mouthwash and instructions on its use. They will subsequently be followed up for up to six months. Every two weeks, participants will fill out a follow-up questionnaire on mouthwash use and sexual activities and self-collect oral rinse sample to be returned by mail.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years old
* Sexually active and have had oral sex in the past month
* Will be residing in Montreal for the next six (6) months after study enrolment

Exclusion Criteria:

* Previous vaccination against HPV
* Previous cancer of the mouth or throat

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  This will be measured by the total number of participants recruited into the study. The investigators intend to recruit 40 participants. Recruitment rate will be calculated as number of participants per month.
Drop-out rate | 1 year
  The proportion of individuals who enrolled into the study but left before the end of the study will be documented.
Adherence rate for mouthwash use | 6 months
  This will be calculated as the proportion of participants who completed the study and complied with the mouthwash use regimen.
Adherence rate for self-sampling | 6 month
  This will be calculated as the proportion of participants who completed the study and complied with the bi-weekly self-sampling procedure
Acceptability of study procedures as assessed by satisfaction on a Visual Analog Scale | 6 months
  Qualitative and quantitative assessment will be used to evaluate participants' experience with the RCT through the follow-up questionnaire and an exit question. Participants will be asked to rate their satisfaction with the study procedure on a scale of 1-10 (10 being the highest satisfaction level). This will focus on level of satisfaction of the participants with mouthwash use around sexual activities and the level of satisfaction of the participants with the biweekly self-sampling.

SECONDARY OUTCOMES:
Mouthwash safety (Pain score) as assessed by the Visual Analog Scale | 6 months
  The mean pain score (for any pain ascribed to the mouthwash e.g., burning mouth, recurrent aphthous stomatitis e.t.c.) measured on the VAS (1-10; 10 being the worst pain) will be recorded.

OTHER OUTCOMES:
Time to oral HPV infection | 6 months
  Time to type-specific oral HPV infection will be recorded for participants with negative type-specific oral HPV status at baseline
Time to oral HPV clearance | 6 months
  Time to type-specific oral HPV clearance will be recorded for participants with positive type-specific oral HPV status at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Nicolau, DDS, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alli BY, Madathil S, Tran SD, Nicolau B. Protocol: carrageenan for the prevention of oral HPV infection - a feasibility randomised clinical trial. BMJ Open. 2023 Jul 27;13(7):e074498. doi: 10.1136/bmjopen-2023-074498. PMID 37500273